CLINICAL TRIAL: NCT01673828
Title: A Double-blind, Placebo-controlled, Randomized Clinical Trial of Allopregnanolone for the Treatment of Traumatic Brain Injury
Brief Title: Allopregnanolone for the Treatment of Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael A. Rogawski, MD, PhD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Michael A. Rogawski, MD, PhD, Principal Invstigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 273147; DR081314 (Other: UC Davis)
Record Dates: First submitted 2012-08-20; First posted 2012-08-28 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Traumatic Brain Injury; Posttraumatic Epilepsy
Keywords: Brain Injuries; Pregnanolone; Epilepsy
MeSH Terms: conditions — Brain Injuries, Traumatic; Epilepsy, Post-Traumatic; Brain Injuries; Epilepsy | interventions — Pregnanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopregnanolone (Experimental): Allopregnanolone injection (intravenous solution) continuous infusion for 5 days
  Interventions: Drug: Allopregnanolone injection
- Placebo (Placebo Comparator): Placebo injection (intravenous solution) continuous infusion for 5 days
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Allopregnanolone injection — Allopregnanolone intravenous solution in 0.9% sodium chloride injection with 6% sulfobutyl ether β-cyclodextrin sodium
  Other Names: 3α,5α-tetrahydroprogesterone; 3α-hydroxy-5α-pregnan-20-one; Product L (allopregnanolone intravenous solution, low dose); Product H (allopregnanolone intravenous solution, high dose)
  Arms: Allopregnanolone
Drug: Placebo injection — Placebo intravenous solution, 0.9% sodium chloride injection with 6% sulfobutyl ether β-cyclodextrin sodium
  Other Names: Product P (placebo)
  Arms: Placebo

SUMMARY:
This study will provide initial data on the safety and effectiveness of allopregnanolone in improving neurobehavioral outcome and reducing mortality in adults with moderate and severe traumatic brain injury.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, dose-finding, two-stage adaptive, clinical trial study comparing allopregnanolone to placebo when administered intravenously for 5 days beginning within 8 hours after injury. Test products to be administered are low and high dose allopregnanolone (Products L and H, respectively) and placebo (Product P) intravenous solutions. The products are administered during a 4-day treatment period followed by a 1-day dose de-escalation period. Stage 1 of the study will assess safety and confirm that dosing with Products L and H achieve the target steady-state plasma concentrations set for each of these products. Dosing will be adjusted in Stage 1, if necessary. Stage 2 will initially allocate subjects equally to Products L, H and P but will then use adaptive randomization to allocate subjects between Products L and H to optimized the probability of yielding a better 3-month Glasgow Outcome Score Extended (GOS-E) score.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking person
* Moderate to severe closed or blunt traumatic brain injury [post resuscitation Glasgow Coma Score (GCS) 3-12 with abnormal head CT scan if GCS is 9-12]
* Less than 8 hours from injury to study initiation
* Able to participate for the full term of the study

Exclusion Criteria:

* Subjects with life expectancy of less than 24 hours
* Isolated epidural hematoma
* Hypoxia (pulse oximetry saturation ≤90% for 15 or more minutes before enrollment)
* Hypotension (systolic blood pressure ≤90 mm Hg on 2 or more reliable measurements before enrollment)
* Cardiopulmonary arrest prior to randomization
* Spinal cord injury with motor deficits
* Bilateral non-reactive pupils with Glasgow Coma Scale 3
* Body weight >120 kg
* Pregnancy
* Active breast or reproductive organ cancer
* Allergy to progesterone
* History of thromboembolic events
* Receipt of activated Factor VII before enrollment
* Any disease that is unstable or which could jeopardize the safety of the subject including severe renal impairment (creatinine clearance <50 ml/min)
* Prisoner/ward of the state
* Known treatment with another investigational drug therapy or procedure within 30 days of injury

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Rogawski, MD, PhD, Principal Investigator — University of California, Davis; JoAnne E Natale, MD, PhD, Study Director — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allopregnanolone | Placebo
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopregnanolone | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (13.1) | 26.2 (13.5) | 28.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
TBI Severity [Count of Participants; unit: Participants] — Moderate=post-resuscitation Glasgow Coma Scale (GCS) within range of 9-12 with abnormal head CT scan. Severe=post-resuscitation GCS within range of 3-8.
  Participants
    Moderate | 2 | 0 | 2
    Severe | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Extended Glasgow Outcome Scale (GOS-E) Score
Description: GOS-E is a global scale for functional outcome that rates patient status into one of 8 levels. The minimum score is 1 and the maximum score is 8. 1 = dead; 2 = vegetative state; 3 = low severe disability; 4 = upper severe disability; 5 = low moderate disability; 6 = upper moderate disability; 7 = low good recovery; 8 = upper good recovery. GOS-E was assessed by 19 question structured interview.
Time Frame: 6 months after injury
Measure: Mean (Standard Deviation); unit: GOS-E Score
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 7 | 6
GOS-E Score | 4.2 (1.9) | 4.3 (1.8)

ADVERSE EVENTS:
Arm/Group | Allopregnanolone | Placebo
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 7/7 | 6/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopregnanolone (N=7) | Placebo (N=6)
Leg compartment syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epidural hematoma (Nervous system disorders) | 0 (0) | 2 (2)
Hemorrhage (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hypotension (Cardiac disorders) | 5 (5) | 3 (3)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Intreased intracranial pressure (Nervous system disorders) | 6 (6) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Brain herniation (transtentorial and uncal) (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopregnanolone (N=7) | Placebo (N=6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Jaundice (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary edema (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 1 | 0 (0)
Conjunctival edema (Eye disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Alcohol withdrawal symptom (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Cerebral hypoperfusion (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Central venous pressure decrease (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QTC interval prolonge (Investigations) | 2 (2) | 4 (4)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0)
Internation normalized ratio increase (Investigations) | 0 (0) | 1 (1)
Diabetes insipidus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypervolemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Craniocerebral injury (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increase (Nervous system disorders) | 6 (6) | 6 (6)
Meningitis (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Spinal epidural hematoma (Nervous system disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 3 (3) | 2 (2)
Drug withdrawal syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonia staphylococcal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eschar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 5 (5) | 3 (3)
Pulmonary embolism/deep vein thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sacrum ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
One subject receiving active treatment died during initial hospitalization; the death was not considered related to the study treatment. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes